CLINICAL TRIAL: NCT01396694
Title: Phase 4 Study of the Influence of Psychological Factors on the Outcomes Following Arthroscopy and Arthroplasty for Temporomandibular Joint Dysfunction
Brief Title: An Evaluation of Psychological Parameters That May Influence the Outcome Following Arthroscopy and Arthroplasty for Temporomandibular Joint Surgery
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Gary F Bouloux MD, DDS, MDSc, FRACDS, FRACDS, PI, Emory University
Other Study IDs: IRB00061869
Record Dates: First submitted 2011-07-08; First posted 2011-07-19 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Psychological Predictors
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- all: All patients requiring arthroscopy or arthroplasty
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaire

SUMMARY:
All patients undergoing arthroscopy or arthroplasty for temporomandibular joint dysfunction will complete a psychological questionnaire prior to surgery. The 3 month outcomes including pain and function will be examined using regression analysis to identify psychological variables that may predict outcomes.

ELIGIBILITY:
Inclusion Criteria:

* require arthroscopy or arthroplasty

Exclusion Criteria:

* age less than 18 yrs
* prior surgery
* unable to give informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18 yrs
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2009-06; Primary Completion 2012-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Pain | 3 months
  Pain will be recorded in a site specific matter (left and right TMJ) using a visual analogue scale

SECONDARY OUTCOMES:
Function | 3 months
  Function will be measured using the jaw function limitation scale which will assess overall jaw and masticatory function with a short well validated questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Emory University, Atlanta, Georgia, United States